CLINICAL TRIAL: NCT05336994
Title: Patterns of Plasma Vitamins and Minerals Following Intake of a Multivitamin/ Mineral Formula Produced by Two Different Manufacturing Processes
Brief Title: Vitamin/Mineral Absorption From Two Different Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 1692409
Record Dates: First submitted 2022-03-24; First posted 2022-04-20 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Healthy Nutrition
Keywords: Minerals; Vitamins; Absorption
MeSH Terms: interventions — Geritol

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive either supplement A or supplement B during the first visit. Five to seven days later, participants will receive the other supplement.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multivitamin/mineral supplement A to B (Experimental): Participants will be randomly assigned to receive Supplement A and after 5-7 days of follow-up, they will receive Supplement B.
  Interventions: Dietary Supplement: Multivitamin/mineral supplement A; Dietary Supplement: Multivitamin/mineral supplement B
- Multivitamin/mineral supplement B to A (Experimental): Participants will be randomly assigned to receive Supplement B and after 5-7 days of follow-up, they will receive Supplement A.
  Interventions: Dietary Supplement: Multivitamin/mineral supplement A; Dietary Supplement: Multivitamin/mineral supplement B

INTERVENTIONS:
Dietary Supplement: Multivitamin/mineral supplement A — Oral administration of Supplement A
Dietary Supplement: Multivitamin/mineral supplement B — Oral administration of Supplement B

SUMMARY:
The objective of this project is to evaluate the postprandial serum and plasma vitamin and mineral levels in healthy adult men and women between 18 and 32 years of age, following a single intake of a multivitamin and mineral supplement processed in two different ways.

DETAILED DESCRIPTION:
Serum or plasma levels of five vitamins and four minerals will be measured at baseline, and 1, 2, 4, and 6 hours after the intake of a multivitamin/mineral supplement processed by two different methods. The two methods involve using either conventional isolated vitamins and minerals blended together to provide approximately 100% of the Daily Value, or using the same amount of vitamins and minerals that have first been processing into liposomal forms before blending.

Participants are required to come for two study visits which are 5 to 7 days apart. Health screening will also be done at Study Visit 1. The order of supplement assignment will be randomized, performed in a double-blind manner.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females 18-32 years of age
* BMI 18.5-32 kg/m2
* Free from disease
* Normal blood levels in the comprehensive metabolic panel, or values slightly out of range as approved by the study physician
* Normal blood pressure (individuals whose average blood pressure is greater than 140/90 will be excluded from the study)
* Suitable vein structure and access for successful placement of an indwelling catheter, as determined by our nurse phlebotomist

Exclusion Criteria:

* Alcohol consumption > 3 drinks/week (i.e., 1 bottle of beer, 1 glass of wine, and 1 shot of hard liquor)
* Smoking
* Vaping or using cannabis in any form
* Using multivitamin/mineral supplements in the past two months
* Currently taking supplements including botanical supplements, probiotics or fiber
* Fruit consumption ≥ 2 cups/day
* Vegetable consumption ≥ 3 cups/day
* Coffee/tea ≥ 3 cups/day
* Chronic/routine high-intensity exercise
* Any chronic health conditions
* Self-reported malabsorption
* Currently taking prescription drugs
* Indications of substance or alcohol abuse within the last 3 years
* Unable to consent

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Assess the serum or plasma levels of five vitamins and four minerals | 6 hours
  Total area-under-the-curve of serum Vitamin A
Assess the serum or plasma levels of five vitamins and four minerals | 6 hours
  Total area-under-the-curve of serum folate
Assess the serum or plasma levels of five vitamins and four minerals | 6 hours
  Total area-under-the-curve of serum Vitamin D
Assess the serum or plasma levels of five vitamins and four minerals | 6 hours
  Total area-under-the-curve of serum Vitamin B-12
Assess the serum or plasma levels of five vitamins and four minerals | 6 hours
  Total area-under-the-curve of plasma Vitamin C
Assess the serum or plasma levels of five vitamins and four minerals | 6 hours
  Total area-under-the-curve of serum zinc
Assess the serum or plasma levels of five vitamins and four minerals | 6 hours
  Total area-under-the-curve of serum iron
Assess the serum or plasma levels of five vitamins and four minerals | 6 hours
  Total area-under-the-curve of serum manganese
Assess the serum or plasma levels of five vitamins and four minerals | 6 hours
  Total area-under-the-curve of serum magnesium

SECONDARY OUTCOMES:
Assess the serum or plasma levels of five vitamins and four minerals | 6 hours
  Maximum serum level of Vitamin A (mg/dL)
Assess the serum or plasma levels of five vitamins and four minerals | 6 hours
  Maximum serum level of folate (mg/dL)
Assess the serum or plasma levels of five vitamins and four minerals | 6 hours
  Maximum serum level of Vitamin D (mg/dL)
Assess the serum or plasma levels of five vitamins and four minerals | 6 hours
  Maximum serum level of Vitamin B-12 (mg/dL)
Assess the serum or plasma levels of five vitamins and four minerals | 6 hours
  Maximum plasma level of Vitamin C (mg/dL)
Assess the serum or plasma levels of five vitamins and four minerals | 6 hours
  Maximum serum level of zinc (mg/dL)
Assess the serum or plasma levels of five vitamins and four minerals | 6 hours
  Maximum serum level of iron (mg/dL)
Assess the serum or plasma levels of five vitamins and four minerals | 6 hours
  Maximum serum level of manganese (mg/dL)
Assess the serum or plasma levels of five vitamins and four minerals | 6 hours
  Maximum serum level of magnesium (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M. Hackman, PhD, Principal Investigator — Research Nutritionist
Locations (1):
- Ragle Human Nutrition Research Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No